CLINICAL TRIAL: NCT04989465
Title: An Open Phase Ⅳ Clinical Trial to Evaluate the Immunity Persistence After Single Dose of 23-valent Pneumococcal Polysaccharide Vaccine
Brief Title: A Clinical Trial of 23-valent Pneumococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-PPV-4001
Record Dates: First submitted 2021-07-25; First posted 2021-08-04 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2021-06

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 450 Participants (including 150 subjects aged 2~17 years, 150 subjects aged18~60 years and 150 subjects aged 61years and older ) received one dose of 23-valent pneumococcal polysaccharide vaccine manufactured by Sinovac Biotech Co., Ltd will be collected venous blood about 3.0~3.5 ml.
  Interventions: Biological: Investigational 23-valent PPV
- Control Group (Placebo Comparator): 150 Participants (including 50 subjects aged 2~17 years, 50 subjects aged18~60 years and 50 subjects aged 61years and older ) received one dose of 23-valent pneumococcal polysaccharide vaccine manufactured by Chengdu Institute of Biological Products will be collected venous blood about 3.0~3.5 ml.
  Interventions: Biological: Control 23-valent PPV

INTERVENTIONS:
Biological: Investigational 23-valent PPV — The investigational vaccine was manufactured by Sinovac Biotech Co., Ltd.25μg each for serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in 0·5 mL of sodium chloride, sodium dihydrogen phosphate and disodium hydrogen phosphate per injection
  Arms: Experimental Group
Biological: Control 23-valent PPV — The control vaccine was manufactured by Chengdu Institute of Biological products Co., Ltd. 25μg each for serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in 0·5 mL of light disodium phenol phosphate, sodium hydrogen phosphate and sodium chloride per injection
  Arms: Control Group

SUMMARY:
This an open phase Ⅳ clinical trial of 23-valent pneumococcal polysaccharide vaccine manufactured by Sinovac Biotech Co., Ltd.The purpose of this study is to evaluate the immunity persistence after single dose of 23-valent pneumococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
This study is an open phase Ⅳ clinical trial to evaluate the immunity persistence after single dose of 23-valent pneumococcal polysaccharide vaccine.The experimental vaccine was manufactured by Sinovac Biotech Co., Ltd,the control vaccine was manufactured by Chengdu Institute of Biological products Co., Ltd..A total of 600 subjects including 450 subjects in the experimental group and 150 subjects in the control group who participated in the second stage of phase Ⅲ clinical trial (PPS)will be enrolled .Based on the age at the time of enrollment in the phase Ⅲ study, there will be 150 participants in each age group (2-17 years old group, 18-60 years old group and ≥61 years old) in the experimental group and 50 participants in each age group in the control group .3.0-3.5ml of venous blood will be collected from all subjects after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in the second stage of phase Ⅲ clinical trial (PPS);
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8-17 years, both subjects and guardians need to sign the informed consent form);
* Proven legal identity.

Exclusion Criteria:

* Have received any pneumococcal vaccine after participating the phase III clinical trial of 23-valent pneumococcal polysaccharide vaccine ;
* History of invasive disease caused by streptococcus pneumoniae after participating the phase III clinical trial of 23-valent pneumococcal polysaccharide vaccine;
* Autoimmune disease or immunodeficiency / immunosuppression was known after participating the phase III clinical trial of 23-valent pneumococcal polysaccharide vaccine;
* History of immunosuppressive therapy after participating the phase III clinical trial of 23-valent pneumococcal polysaccharide vaccine;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index 1-geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody | From the beginning of the vaccination to 28 days after the full vaccination
  Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody at day 28 after the full vaccination in all subjects
Immunogenicity index 2-geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody | From the beginning of the vaccination to 6 years after the full vaccination
  Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody in 6 years after the full vaccination in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Lili Huang, Master, Principal Investigator — Henan Provincial Center for Disease Prevention and Control
Locations (1):
- Kaifeng County Center for Disease Control and Prevention, Kaifeng, Henan, China